CLINICAL TRIAL: NCT00344266
Title: Gene Expression and Release of Inflammatory Mediators in Overweight Subjects Before and After Weight Loss
Brief Title: Gene Expression and Inflammation in Overweight Subjects
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 060183; 06-DK-0183
Record Dates: First submitted 2006-06-23; First posted 2006-06-26 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2018-06-26

CONDITIONS: Obesity; Inflammation; Nutrition Therapy
Keywords: Obesity; Adipose Tissue; Microarrays; Cytokines; Eicosanoids; Gene Expression; Adipokines; Inflammation; Weight Loss; Lipid Products
MeSH Terms: conditions — Obesity; Inflammation; Weight Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
This study will look at gene expression (whether particular sets of genes are activated ["turned on"] or deactivated ["turned off"]) in overweight people as compared to non-overweight individuals. It will also investigate the potential role of inflammatory and protective substances that are produced naturally by the body within fat tissue. Findings from the study may lead to the development of ways to predict who will respond best to diet therapy.

Healthy individuals between 25 and 45 years of age may be eligible for this study. Overweight subjects must have a BMI of 25 to 40, and non-overweight control subjects a BMI of 19 to 24.9. Candidates are screened with a medical history, physical examination, blood tests and electrocardiogram (EKG). They are instructed to record their dietary intake for a 3-day period and to collect their urine for a 24-hour interval.

Participants have their food records reviewed a week after the screening visit. They are then scheduled for an overnight admission to the Clinical Center. Non-overweight subjects have one or two inpatient stays; overweight subjects have six inpatient stays plus frequent nutrition counseling sessions. During the 2-day hospital admissions, the following studies are performed:

* DEXA scan to determine the percentage of body fat tissue. The subject lies on a table for about 15 to 60 minutes while the body composition is measured with very low-dose x-rays.
* Single-slice CT scan to compare the amount of fat tissue under the skin with that in the abdomen. The subject lies on a table for about 5 to 10 minutes while the CT scanner measures body composition with very low-dose x-rays.
* Subcutaneous fat microdialysis to investigate how weight loss affects the activity of fat tissue. A small tube (catheter) is placed into the fat tissue under the skin of the abdomen after numbing the skin with a local anesthetic. Fluid samples are collected through the tube. The procedure lasts overnight. In five non-overweight controls, a small amount of a substance called leukotriene B4 is put into their fat tissue to help adjust the instruments used in the study.
* Air-displacement plethysmography to measure body composition. Subjects wear close-fitting clothing and enter a small capsule called a Bod-Pod. They breathe normally in the capsule while their body fat composition is studied.
* Blood tests. Blood samples are drawn to analyze thyroid hormones, lipids, glucose, electrolytes, clotting factors, kidney function, red cells and DNA.
* Euglycemic-hyperinsulinemic clamp to measure the effects of insulin in the body and to derive an index of insulin-sensitivity. Catheters are placed in a vein in an arm and in a vein in the hand on the other side of the body. Insulin and glucose are infused through the catheter in the arm, and blood samples are drawn from the catheter in the hand every 5 minutes to measure glucose levels. The test lasts about 2 hours.
* Subcutaneous fat biopsy to find out how weight loss affects fat tissue characteristics, gene regulation and the ability to store glucose. A small sample of fat tissue is obtained from the skin of the abdomen after numbing the area with an anesthetic.
* Nutrition counseling for overweight subjects. A nutritionist reviews the food record and designs a personalized diet for each participant.
* Weight loss intervention for overweight subjects. In addition to individual nutritional counseling, group sessions are provided every 2 weeks during the first 3 months of the study and then every month.

DETAILED DESCRIPTION:
Obesity is a global public health problem of epidemic proportions. It is the source of considerable morbidity and early mortality in the U.S. and is associated with increased risk of diabetes, hypertension, cardiovascular disease, and cancer.

In recent years, new and evolving concepts have emerged regarding obesity as a chronic endocrine disorder of inflammation. Moreover, a growing body of evidence indicates that obesity alters the profile of a constellation of genes and that some changes in biomarkers of inflammation and gene expression can be reversed by weight loss.

In this clinical protocol, we propose to test the idea that a particular set of genes is activated (or deactivated) in Overweight Subjects using standard microarray techniques on samples of subcutaneous adipose tissue derived from biopsies. In addition, we will study the local adipose tissue microenvironment by means of microdialysis. The role of a number of adipokines, inflammatory mediators/cytokines, and novel lipid products will be analyzed using sensitive Liquid Chromatography-Mass Spectrometry and ELISA methods.

The study design incorporates two basic objectives:

1. Comparison of Non-Overweight Controls vs. Overweight Subjects at Baseline and
2. Correlation of changes in Overweight patients over time as they lose weight through a calorie-restricted diet.

To these ends, 30 Non-Overweight Controls (BMI 19.0 24.9) and 80 Overweight Subjects (BMI 25.0 45.0) will be enrolled. Baseline studies, to be obtained on all participants include: blood tests, anthropometric indices, body composition by air-displacement plethysmography, indirect calorimetry, intravenous glucose tolerance test as an index of insulin sensitivity, subcutaneous adipose tissue microdialysis, and subcutaneous adipose tissue biopsy. These procedures will require an overnight hospital admission to the Clinical Center. Overweight Subjects will then be prescribed a calorie-restricted diet and followed for one year. They will undergo repeat studies at regular, 3-month intervals to assess serial changes in the various parameters and to provide correlative data with the degree and rate of weight loss achieved.

Taken together, these studies should shed light and provide fundamental insights into the nature of the altered gene expression and release of inflammatory cytokines and other mediators that characterize the overweight state and the dynamic series of events that take place when dietary intervention leads to weight loss. It is anticipated that a number of these changes will relate to macrophages and known inflammatory markers though doubtless there are other important leads yet to be discovered. Thus, our hope is that such studies will ultimately lead to the identification of novel genes that underlie the important metabolic derangements associated with obesity and their response to different treatment modalities.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age 25-45 years, male or female
* BMI 25.0-45.0 kg/m(2) for Overweight Subjects and 19.0-24.9 kg/m(2) for Non-Overweight Controls
* Healthy, as determined by medical history and laboratory tests
* Written informed consent

EXCLUSION CRITERIA:

* BMI less than 19.0 or greater than 45.0 kg/m(2)
* History or symptoms compatible with cardiovascular disease, including arrhythmias and syncopal episodes, or use of prescription medications for heart conditions, strokes, or peripheral vascular disease
* Allergy to lidocaine
* Pregnancy or breastfeeding
* Menopause or peri-menopausal period (FSH greater than 15 mIU/ml)
* Use of hormonal contraceptives or estrogen replacement therapy
* Alcohol (more than 2 drinks per day or CAGE greater than 2 questions and/or current/regular use of drugs such as amphetamines, cocaine, heroin, or marijuana
* Current use of tobacco products (smoking or chewing)
* History of Diabetes Mellitus, either type 1 or 2, or Fasting Glucose greater than 126 mg/dl
* Use of cholesterol- or lipid-lowering drugs, or fasting serum lipids in range requiring medication per Adult Treatment Panel III recommendations of the National Cholesterol Education Program
* Liver disease or ALT serum level greater than two-fold above the laboratory reference standard
* Renal insufficiency or estimated creatinine clearance less than or equal to 50 ml/min
* Current use of medications, dietary supplements (including fish oils), or alternative therapies known to alter thyroid function with the exception of occasional use of NSAIDs (3 tablets/week maximum) and Benzodiazepines; use of NSAIDs in the 10 days preceding the hospital admissions
* Current history, symptoms, or behavior compatible with psychiatric disorders or therapy with psychotropic medications that would be incompatible with safe and successful participation in this study
* History of drug or alcohol abuse within the last 5 years; current use of drugs or alcohol
* Keloid formation (relative to subcutaneous adipose tissue biopsies)
* Hypo- or hyperthyroidism (TSH greater than or equal to 10; less than or equal to 0.1 mIU/L)
* Blood pressure greater than 160/95 mm Hg or use of prescription medications for treatment of hypertension
* Cushing Syndrome

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 144 (Actual)
Dates: Start 2006-06-19; Study Completion 2018-06-26

PRIMARY OUTCOMES:
Adipokines/cytokines in adipose tissue | End of study
Gene expression in adipose tissue | End of study

CONTACTS AND LOCATIONS:
Overall Officials: Kong Y Chen, Ph.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Arita M, Clish CB, Serhan CN. The contributions of aspirin and microbial oxygenase to the biosynthesis of anti-inflammatory resolvins: novel oxygenase products from omega-3 polyunsaturated fatty acids. Biochem Biophys Res Commun. 2005 Dec 9;338(1):149-57. doi: 10.1016/j.bbrc.2005.07.181. Epub 2005 Aug 10. PMID 16112645
- [Background] Brown RL, Leonard T, Saunders LA, Papasouliotis O. A two-item conjoint screen for alcohol and other drug problems. J Am Board Fam Pract. 2001 Mar-Apr;14(2):95-106. PMID 11314930
- [Background] Arner P, Bolinder J. Microdialysis of adipose tissue. J Intern Med. 1991 Oct;230(4):381-6. doi: 10.1111/j.1365-2796.1991.tb00461.x. PMID 1919434
- [Derived] Agnihothri RV, Courville AB, Linderman JD, Smith S, Brychta R, Remaley A, Chen KY, Simchowitz L, Celi FS. Moderate weight loss is sufficient to affect thyroid hormone homeostasis and inhibit its peripheral conversion. Thyroid. 2014 Jan;24(1):19-26. doi: 10.1089/thy.2013.0055. PMID 23902316